CLINICAL TRIAL: NCT05741957
Title: Examining the Optimal Exercise Frequency for Alleviating Liver Fat in Centrally Obese Adults With Non-Alcoholic Fatty Liver Disease (NAFLD): A Comparative Randomized Controlled Trial
Brief Title: Optimal Exercise Frequency to Reduce Liver Fat in Centrally Obese Adults With Non-Alcoholic Fatty Liver Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Associate Professor and Division Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKU-NFF
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
Keywords: Non-Alcoholic Fatty Liver Disease; Overweight; Central Obesity; Obesity; Adults; Aerobic Exercise; Exercise Frequency
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Overweight; Obesity, Abdominal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Once-a-week Exercise (Experimental): Once-a-week vigorous-intensity exercise for 4 months.
  Interventions: Behavioral: Once-a-week Exercise
- Thrice-a-week Exercise (Experimental): Thrice-a-week vigorous-intensity exercise for 4 months.
  Interventions: Behavioral: Thrice-a-week Exercise
- Usual Care Control (Other): Bi-weekly health education for 4 months.
  Interventions: Other: Usual Care Control

INTERVENTIONS:
Behavioral: Once-a-week Exercise — Participants in this group will participate in a supervised treadmill exercise program delivered by certified fitness instructors. The prescribed program will involve one session weekly for 4 months, and the duration of vigorous-intensity treadmill exercise per session will be 75 min. Participants will exercise with an exercising heart rate at 6-7 metabolic equivalents (METs). Health information provided to the usual care control group will be made available to the participants in this group.
  Arms: Once-a-week Exercise
Behavioral: Thrice-a-week Exercise — Participants in this group will participate in a supervised treadmill exercise program delivered by certified fitness instructors. The prescribed program will involve three sessions weekly for 4 months, and the duration of vigorous-intensity treadmill exercise per session will be 25 min. Participants will exercise with an exercising heart rate at 6-7 METs. Health information provided to the usual care control group will be made available to the participants in this group.
  Arms: Thrice-a-week Exercise
Other: Usual Care Control — Participants in this group will receive health education delivered by research personnel. This program will consist of eight two-hour bi-weekly sessions covering major health issues relating to general health and NAFLD, such as non-communicable diseases, infectious diseases, and a healthy lifestyle.
  Arms: Usual Care Control

SUMMARY:
This study aims to examine the comparative effectiveness of different exercise frequencies (once-a-week vs. thrice-a-week) for reducing liver fat in centrally obese adults with non-alcoholic fatty liver disease (NAFLD), with weekly exercise volumes aligned with the World Health Organization's physical activity recommendations.

DETAILED DESCRIPTION:
This study is a three-arm randomized controlled trial. Participants will be randomly allocated to the once-a-week exercise group, thrice-a-week exercise group, or usual care control group. The exercise intervention groups will receive once-a-week or thrice-a-week exercise (with matched weekly exercise volumes). The usual care control group will receive general health education. All interventions will last for 4 months. Outcome measures will be examined at baseline, 4 months (post-intervention), and 10 months (6-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Cantonese, Mandarin, or English speaking Chinese;
2. Aged 18-69;
3. Male or female;
4. Centrally obese according to the Asian-specific cut-off (waist circumference ≥90 cm for males; ≥80 cm for females) and with BMI ≥23;
5. With NAFLD (defined as >5% intrahepatic triglycerides assessed by 1H-MRS);
6. Willing to participate in exercise training to improve NAFLD.

Exclusion Criteria:

1. Regular exercise training (>3 sessions of >60 min of moderate-intensity exercise training weekly) in the past 6 months;
2. Medical history of cardiovascular disease, chronic pulmonary or kidney disease, heart failure, cancer, and/or liver disease except NAFLD;
3. Somatic conditions that limit exercise participation (e.g., limb loss);
4. Impaired mobility due to chronic disease (e.g., chronic arthritis/osteoarthritis, neurological, musculoskeletal, and autoimmune diseases);
5. Daily smoking habit;
6. Excess alcohol consumption (daily ≥20 g of alcohol for men and ≥10 g for women) in the past 1 year;
7. Consumption of certain drugs (e.g., tamoxifen and estrogen) known to be secondary causes of steatosis;
8. Surgery, therapy, or medication for obesity or weight loss in the past 6 months (e.g., gastric bypass, gastric band, sleeve gastrectomy, gastric reduction duodenal switch, or dietitian-prescribed dietary program);
9. Physical changes that considerably affect body composition and weight (e.g., anorexia nervosa, bulimia nervosa, prolonged gastrointestinal and digestive disorders) during the study period.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Liver Fat | Baseline and 4 months (post-intervention)
  Intrahepatic triglycerides will be assessed using proton magnetic resonance spectroscopy (1H-MRS) in a 3×3×3 cm voxel.

SECONDARY OUTCOMES:
Change in Liver Fat | Baseline and 10 months (follow-up)
  Intrahepatic triglycerides will be assessed using 1H-MRS in a 3×3×3 cm voxel.
Change in Abdominal Visceral Fat | Baseline, 4 months (post-intervention), and 10 months (follow-up)
  Abdominal visceral fat will be assessed using magnetic resonance imaging (MRI).
Change in Body Fat | Baseline, 4 months (post-intervention), and 10 months (follow-up)
  Total body fat mass will be assessed using dual-energy x-ray absorptiometry (DXA).
Change in Body Mass Index | Baseline, 4 months (post-intervention), and 10 months (follow-up)
  Weight and height will be assessed using a calibrated electronic digital weighing scale and a stadiometer, respectively.
Change in Waist Circumference | Baseline, 4 months (post-intervention), and 10 months (follow-up)
  Waist circumference will be assessed using an inelastic measuring tape to the nearest 0.1 cm on bare skin.
Change in Maximal Oxygen Consumption | Baseline, 4 months (post-intervention), and 10 months (follow-up)
  Maximal oxygen consumption will be assessed using the modified Bruce protocol.
Change in Physical Component Summary Score of the 12-Item Short-Form Health Survey | Baseline, 4 months (post-intervention), and 10 months (follow-up)
  Physical health-related quality of life will be assessed using the Physical Component Summary scale of the 12-Item Short-Form Health Survey (SF-12). Scores on the scale range from 0 to 100, with higher scores indicating better physical health-related quality of life.
Change in Mental Component Summary Score of the 12-Item Short-Form Health Survey | Baseline, 4 months (post-intervention), and 10 months (follow-up)
  Mental health-related quality of life will be assessed using the Mental Component Summary scale of the 12-Item Short-Form Health Survey (SF-12). Scores on the scale range from 0 to 100, with higher scores indicating better mental health-related quality of life.
Number of Adverse Events | Baseline, 4 months (post-intervention), and 10 months (follow-up)
  Adverse events related or unrelated to the intervention will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Parco M. Siu, PhD, Principal Investigator — LKS Faculty of Medicine, The University of Hong Kong
Locations (1):
- LKS Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants that underlie the results reported in this trial, after de-identification including text, tables, figures, and appendices, as well as study protocol and statistical analysis plan, will be shared after 3 months of study publication. Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years following the publication of the article.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.